CLINICAL TRIAL: NCT07385677
Title: Comparing the Effectiveness of the 'Think in Nerve Length and Layers' (TINLL) Approach to Traditional Treatment for Patients With Lateral Elbow Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Victoria Priganc, Associate Professor, University of Vermont
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003117
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Lateral Elbow Tendinopathy (Tennis Elbow)
Keywords: lateral elbow pain; radial nerve
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TINLL (Experimental): * radial head mobilization
  * biceps tendon mobilization with movement to address joint alignment, neural tension, and the superficial sensory nervous system.
  * elastic tape cross fiber inhibition 50% stretch over distal biceps
  * elastic tape radial head stabilization with 80% stretch
  * biceps stretching/lengthening
  * pectoralis major stretching
  * scapular strengthening
  * triceps and supinator strengthening
  * ergonomic strategies
  Interventions: Other: TINLL techniques for relieving radial nerve tension
- Traditional (Active Comparator): * stretching of the wrist extensors
  * isometric, concentric, and/or eccentric strengthening of the finger extensors, wrist extensors, pronator, and supinator muscles
  * elbow joint manipulation or mobilization (such as mobilization with movement (MWM) as developed by Mulligan)
  * soft tissue mobilization techniques to the forearm muscles
  * instrument-assisted soft tissue mobilization (IASTM) to the forearm muscles
  * rigid taping techniques and elastic taping application as part of a multimodal treatment program focused on common extensors
  * ergonomic strategies
  * transcutaneous electrical nerve stimulation (TENS)
  * wrist orthosis/splinting
  Interventions: Other: Traditional techniques to stretch and strengthen muscles

INTERVENTIONS:
Other: TINLL techniques for relieving radial nerve tension — 1x/week for 4-6 weeks or less if patient responds well to the treatment
  Arms: TINLL
Other: Traditional techniques to stretch and strengthen muscles — 1x/week for 4-6 weeks unless patients responds well to treatment
  Arms: Traditional

SUMMARY:
Lateral elbow pain can significantly limit people's ability to do the activities they want or need to do. We want to explore if one treatment technique is better than another for people with lateral elbow pain.

You will be placed in a traditional treatment group or in a non-traditional treatment group. Your placement in the group will depend on past treatments you have had for this pain.

Before you start treatment, you will be given four tests: 1) a grip strength test, 2) a pinch test, 3) a pain level survey, and 4) a functional survey. These four tests will take no longer than 15 minutes to complete. These four tests are common tests given to people with elbow pain. You will be given these four tests:

* At the beginning, before you start treatment
* At 2-weeks
* At 4-weeks
* At the end of your treatment

Traditional treatment group: You will receive treatment 1x/week for 4-6 weeks. The traditional treatment group will consist of the following treatments:

* stretching and strengthening of the wrist extensors
* soft tissue work to the forearm muscles
* joint mobilization at the elbow
* rigid and elastic taping with focus on the wrist extensor muscles
* ergonomic strategies
* transcutaneous electrical nerve stimulation (TENS)
* wrist splinting

Non-traditional (TINLL) treatment group: You will receive treatment 1x/every 1-2-weeks for 4-6 weeks. The non-traditional (TINLL) treatment group will consist of the following treatments:

* joint and tendon mobilization at the elbow
* elastic tape for muscles and nerves
* stretching/strengthening of the muscles at the elbow and upper arm
* ergonomic strategies

DETAILED DESCRIPTION:
Upon referral for lateral elbow pain, two schedulers will look at the referral and consult with the study co-investigators to decide what group they should be assigned to based on past medical treatment for lateral elbow pain. The schedulers will have a script they read over the phone to the patients. This will be part of the usual call. At this point, patients do not need to decide whether or not to participate; they are just introduced to the study. Upon arrival for their appointment, the scheduler will introduce the study again to the patient and the patient will be given the opportunity to watch a short video on an approved IPad. This closed-captioned video will provide details of the study and patients will watch the video in a treatment room. After watching the video, the co-investigators will review the consent form and ask the participant if they have any questions. Those subjects that agree to participate will sign the consent form, thus consenting to participate. Those subjects who do not agree to participate will still receive treatment.

Once consent is obtained, subjects will be assigned to either the TINLL group or the traditional treatment and given a research ID number. Once assigned to a group, the therapist in charge of that group will perform the following assessments at the initial visit: numerical rating scale for pain (NRS), patient-rated tennis elbow evaluation (PRTEE), one pain free grip strength with extended elbow and pronated forearm (strength number recorded), and one 3-jaw pinch max effort (pain level and strength number recorded). Regardless of group assignment, all subjects will undergo these assessments at the initial visit. Following the assessments, subjects will begin either the TINLL or the traditional treatment group. Subjects will be assessed at the initial visit, 2-week visit, and 4-week visit and the same assessments will be administered by the same therapist. After the 4-week visit, subjects can opt to switch groups if they choose to do so. These visits described below are regular standard of care intervals. If a subject requires additional visits beyond what is listed below, the subject will be excluded from the study and will receive needed care and billed according to standard practices.

Treatment for the TINLL group will be 1x every 1-2-weeks for 4-6 weeks and consists of a combination of the following depending on the patient:

* radial head mobilization
* biceps tendon mobilization with movement to address joint alignment, neural tension, and the superficial sensory nervous system.
* elastic tape cross fiber inhibition 50% stretch over distal biceps
* elastic tape radial head stabilization with 80% stretch
* biceps stretching/lengthening
* pectoralis major stretching
* scapular strengthening
* triceps and supinator strengthening
* ergonomic strategies

Additional treatments may be considered. These include:

* techniques for relieving radial nerve tension (instrument-assisted soft tissue mobilization (IASTM), silicone cup gliding)
* radial nerve taping from dorsal thenar muscle to C7 on stretch (10%).

The home exercise program for this group includes biceps inhibition tape, radial head stabilization tape, and isometric strengthening triceps/supination (dosing = 1-2 sets/day for 8 reps).

Treatment for the traditional treatment group will be 1x every week for 4-6 weeks and will consist of a combination of the following depending on the patient:

* stretching of the wrist extensors
* isometric, concentric, and/or eccentric strengthening of the finger extensors, wrist extensors, pronator, and supinator muscles
* elbow joint manipulation or mobilization (such as mobilization with movement (MWM) as developed by Mulligan)
* soft tissue mobilization techniques to the forearm muscles
* instrument-assisted soft tissue mobilization (IASTM) to the forearm muscles
* rigid taping techniques and elastic taping application as part of a multimodal treatment program focused on common extensors
* ergonomic strategies
* transcutaneous electrical nerve stimulation (TENS)
* wrist orthosis/splinting
* The home exercise program for this group includes extrinsic stretches for wrist extensors (3 reps, 30 sec holds, 1 time/day) and strengthening (dosing = 3 sets of 15 repetitions 1x/day)

Following 1-month of treatment in either group, subjects will be given the opportunity to switch groups.

6-mo following treatment, subjects will be contacted via phone and asked follow-up questions related pain, function (via the PRTEE), use of taping, and use of home exercises.

ELIGIBILITY:
Inclusion Criteria:

* understanding of English language; adults 18 years of age or older
* referral for lateral sided elbow pain or lateral epicondylitis
* subjects positive on one of the following (tenderness over lateral epicondyle with palpation
* pain with stretch of long wrist extensors
* pain with resisted wrist or middle finger extension)

Exclusion Criteria:

* subjects unable to cognitively follow directions
* have a legally-mandated reporter
* subjects scheduled for surgery, or post-up surgical patients
* subjects with carpal tunnel syndrome, cubital tunnel syndrome/medial elbow pain,
* subjects who received Platelet-Rich Plasma (PRP) or percutaneous needle tenotomy (PNT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Patient rated tennis elbow evaluation (PRTEE) | Day 1, 2-week appointment, 4-week appointment
  15-item, self-report questionnaire designed to measure pain and disability in patients with lateral elbow tendinopathy (tennis elbow).
pain-free grip strength | Day 1, 2-week appointment, 4-week appointment
  pain-free grip strength using Jamar dynamometer
numeric rating scale for pain | Day 1, 2-week appointment, 4-week appointment
  pain scale

SECONDARY OUTCOMES:
3-jaw pinch | Day 1, 2-week appointment, 4-week appointment
  pinch measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedica and Rehabilitation Center - Occupational Therapy/Hand Therapy, University of Vermont Medical Center, South Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared via presentations and/or publications.

REFERENCES:
- [Background] Taylor A, Wolff AL. The forgotten radial nerve: A conceptual framework for treatment of lateral elbow pain. J Hand Ther. 2021 Apr-Jun;34(2):323-329. doi: 10.1016/j.jht.2021.05.009. Epub 2021 Jun 27. PMID 34193382
- [Background] Lucado AM, Day JM, Vincent JI, MacDermid JC, Fedorczyk J, Grewal R, Martin RL. Lateral Elbow Pain and Muscle Function Impairments. J Orthop Sports Phys Ther. 2022 Dec;52(12):CPG1-CPG111. doi: 10.2519/jospt.2022.0302. PMID 36453071
- [Background] Degen RM, Conti MS, Camp CL, Altchek DW, Dines JS, Werner BC. Epidemiology and Disease Burden of Lateral Epicondylitis in the USA: Analysis of 85,318 Patients. HSS J. 2018 Feb;14(1):9-14. doi: 10.1007/s11420-017-9559-3. Epub 2017 Jun 5. PMID 29398988